CLINICAL TRIAL: NCT02989285
Title: The Identification and Quantification of HIV CNS Latency Biomarkers
Brief Title: Identification and Quantification of HIV CNS Latency Biomarkers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St Vincent's Hospital, Sydney (Other)
Responsible Party: Principal Investigator, Bruce Brew, Professor, St Vincent's Hospital, Sydney
Other Study IDs: 15/277; APP1105808 (Other Grant/Funding Number: NHMRC)
Record Dates: First submitted 2016-07-06; First posted 2016-12-12 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: HIV; HIV-associated Neurocognitive Disorder (HAND)
Keywords: HIV; HIV-associated neurocognitive disorder (HAND); Neurology; Latent HIV; HIV Reservoirs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cerebrospinal fluid and bloods
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- HIV+ cognitively impaired (HAND): Participants will be assessed based on their performance on the neuropsychological test battery at study entry. HAND status will be diagnosed per FRASCATI research criteria and this will determine which study cohort they are allocated to. Participants will continue to receive their standard of care treatment during the study period.
- HIV+ cognitively normal (no-HAND): Participants will be assessed based on their performance on the neuropsychological test battery at study entry. HAND status will be diagnosed per FRASCATI research criteria and this will determine which study cohort they are allocated to. Participants will continue to receive their standard of care treatment during the study period.

SUMMARY:
Human Immunodeficiency Virus (HIV) remains in infected patients receiving highly active antiretroviral therapy (HAART) for many years. Stopping HAART usually leads to re-emergence of small reservoirs of latent (inactive) HIV that reside inside certain types of infected cells, that can replicate and cause a full HIV infection. Chronic HIV infection also leads to long-term immune activation which is associated with higher incidence of serious non-AIDS events including cardiovascular disease and cancers. Thus HIV+ patients must remain on HAART indefinitely or replication-competent latent HIV reservoirs must be eradicated.

The central nervous system (CNS) is a sanctuary site for latent HIV. For example, HIV-associated neurocognitive disorders (HAND) develop and persist in about 40% of HIV+ persons despite long-term HAART and viral suppression in blood and cerebrospinal fluid (CSF). Continued CSF immune activation is also frequently observed despite viral suppression. Both of these are likely to indicate ongoing low-level HIV replication in the CNS.

Several strategies to eradicate latent HIV are being explored. One of these, known as "shock and kill" involves "awakening" latent HIV and inducing replication to make it more susceptible to host immune responses and HAART. However, there are several major caveats to its application in the CNS such as the risk of triggering a serious immunoinflammatory response (e.g., meningoencephalitis) that cannot be easily controlled by HAART. Other eradication strategies may also be problematic given that many latency-reversing agents have limited penetration of the blood brain barrier and limited efficacy in astrocyte cells. To improve the effectiveness of new eradication therapies it will be crucial to develop better methods to identify and quantify latent HIV reservoir sites with greater precision.

To identify potential HIV latency biomarkers in the CNS, the investigators will study HIV+ patients stable on HAART and virally-suppressed in blood and CSF over 24 months. Because such a marker should be associated with HAND or its development without changing significantly with HAND progression, half of the sample will have HAND at study entry and half will not. Patients will undergo neuropsychological testing and give blood and CSF samples every 6 months to identify candidate biomarkers and track them prospectively against HAND development and progression. MRI brain scan will also occur at study entry and after 24 months.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* Aged >18 years
* On HAART with viral load suppression (<50 copies / ml) in both plasma and CSF for at least 6 months
* Able to provide informed consent

Exclusion Criteria:

* Non-HIV related neurological disorder or active CNS opportunistic infection as assessed by full blood count, electrolytes, creatinine, glucose, liver function tests, venereal disease reaction level (VDRL), MRI brain scan and CSF analyses for cell count, protein, glucose, culture, VDRL and cryptococcal antigen
* Psychiatric disorders on the psychotic axis, current major depression, current substance use disorder and/or 12 month history of severe substance use disorder
* Active Hepatitis C co-infection
* History of severe traumatic brain injury (post-traumatic amnesia (PTA) duration>1 day) or loss of consciousness > 30 minutes from other cause (e.g., hypoxic brain injury)
* Non-proficient in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV+ patients who are stable on HAART and have achieved viral suppression in blood and CSF who attend outpatient hospital and primary care clinics.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2016-07; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change in Mean CSF BCL11b levels at 24 months (latency burden biomarker) | Baseline and 24 months
  BCL11b is a C2H5 zinc-finger DNA binding protein that is expressed in the brain and immune system and inhibits HIV gene transcription by recruiting chromatin modifiers and establishing a heterochromatic environment in HIV-infected microglia. It is a promising candidate biomarker for latent HIV infection in the brain. Change in CSF BCL11b levels from baseline at 24 months will be reported. BCL11b will also be tracked against HAND development/progression at each visit to determine its suitability as a marker of latent HIV reservoir size.
Change in Mean Level of 1H-MRS Myo-Inositol in Frontal White Matter at 24 months (latency burden biomarker) | Baseline and 24 months
  Myo-Inositol (mIo) is a brain metabolic marker measured by 1H-Magnetic Resonance Spectroscopy (MRS) that is thought to reflect astroglia and microglia activation in cognitively-impaired individuals. The finding that mIo in the frontal white matter is elevated in HIV+ individuals and remains elevated with HAND progression while other metabolite levels fluctuate, supports its possibility as a HIV latency biomarker. Change in 1H-MRS mIo levels in the FWM from baseline at 24 months will be reported. mIo will also be tracked against HAND development/progression to determine its suitability as a marker of latent HIV reservoir size.
Change in Mean CSF HIV RNA by Single Copy Assay at 24 months (latency significance biomarker) | Baseline and 24 months
  Single copy assay (SCA) of CSF HIV RNA will allow for precise detection of intermittent HIV brain infection productivity at low levels. This assay is highly sensitive and can measure levels of HIV RNA as low as 0.3 copies per ml. Change in CSF HIV RNA levels from baseline at 24 months will be reported. Detectability of CSF HIV RNA by SCA is related to increased risk of HAND development in asymptomatic patients suggesting that it may reflect a marker of latent HIV reservoir significance (i.e., the potential for latent HIV replication that is not defective). Such a marker would be expected to change with incident HAND/progression while having no relationship to latency burden biomarkers (i.e., BCL11b).
Change in Mean CSF HIV tat at 24 months (latency significance biomarker) | Baseline and 24 months
  Tat is a post-transcriptional regulatory protein that promotes inflammation and enhances the effectiveness of HIV transcription to neighbouring cells. Therefore it may act as a latency significance biomarker. Change in CSF HIV tat levels from baseline at 24 months will be reported. HIV tat will be tracked against HAND development/progression and as a latency significance biomarker would be expected to change with incident HAND/progression while having no relationship to latency burden biomarkers (i.e., BCL11b).
Change in Mean CSF neopterin at 24 months (latency significance biomarker) | Baseline and 24 months
  Neopterin is an immune activation biomarker that is elevated in almost all persons with HAND on antiretroviral medication and in some without HAND, supporting its possible role as a latency significance marker. Change in CSF neopterin levels from baseline at 24 months will be reported. CSF neopterin will be tracked against HAND development/progression and as a latency significance biomarker would be expected to change with incident HAND/progression while having no relationship to latency burden biomarkers (i.e., BCL11b).
Change in Mean CSF MCP-1 at 24 months (latency significance biomarker) | Baseline and 24 months
  CSF MCP-1 is an immune activation biomarker that has been found to correlate with change in HAND status. Therefore it may be a latency significance marker. Change in CSF MCP-1 levels from baseline at 24 months will be reported. CSF MCP-1 will be tracked against HAND development/progression and as a latency significance biomarker would be expected to change with incident HAND/progression while having no relationship to latency burden biomarkers (i.e., BCL11b).
Change in Mean CSF NFL at 24 months (latency significance biomarker) | Baseline and 24 Months
  CSF NFL is a marker of neuronal injury. It has been shown to correlate with HAND severity and predict its development, suggesting that it is likely to serve as a latency significance biomarker. Change in CSF NFL levels from baseline at 24 months will be reported. CSF NFL will be tracked against HAND development/progression and as a latency significance biomarker would be expected to change with incident HAND/progression while having no relationship to latency burden biomarkers (i.e., BCL11b).

SECONDARY OUTCOMES:
Correlation between CSF HIV tat, neurocognitive global deficit score, neopterin, and MCP-1 at 24 months | Baseline and 24 months
  Cumulative levels of HIV tat in CSF will be quantified from baseline to 24 months as per primary outcome #4. They will then be correlated against HAND development/progression as quantified by neurocognitive global deficit score (GDS), and levels of inflammatory markers neopterin and MCP-1.
Role of Pre-Integration-Targeting HAART in Reducing HIV Latency Burden | Baseline and 6 months, 12 months, 18 months, and 24 months
  Cumulative HAART history will be recorded and scored as follows: drugs that target the pre-integration/integration phase of HIV replication will be given a score of 1; other drugs will be given a score of 0. Total scores will then be correlated with CSF BCL11b levels and any other CNS latency marker that is identified during primary outcome analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce J Brew, MBBS, MD, Principal Investigator — St Vincent's Hospital, Sydney
Locations (1):
- St Vincent's Hospital, Sydney, Darlinghurst, New South Wales, Australia